CLINICAL TRIAL: NCT01151618
Title: Evaluating Forced Oscillation Technique (FOT) in Abolishing Flow Limitation in Patients With Stable Chronic Pulmonary Disease (COPD)
Brief Title: Evaluating Forced Oscillation Technique (FOT) in Abolishing Flow Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRC-1018-FOTVal-SS
Record Dates: First submitted 2010-06-21; First posted 2010-06-28 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respironics Synchrony ventilator (Non Invasive Ventilation) (Experimental): Non Invasive Ventilation using forced oscillation technique (FOT)
  Interventions: Device: Respironics Synchrony ventilator (Non Invasive Ventilation)

INTERVENTIONS:
Device: Respironics Synchrony ventilator (Non Invasive Ventilation) — Non Invasive Ventilation using forced oscillation technique (FOT)

SUMMARY:
To validate the capability of the Respironics Synchrony ventilator to properly detect Expiratory Flow Limitation (EFL) as compared to the gold standard method of detecting EFL via the Mead and Wittenberger technique.

DETAILED DESCRIPTION:
Positive end expiratory pressure (PEEP) is used in COPD patients to counteract the intrinsic PEEP (PEEPi), which represents the end expiratory recoil pressure of the total respiratory system due to the presence of dynamic hyperinflation (DH).

DH commonly occurs in COPD, where the presence of expiratory flow-limitation (EFL) requires the patient to breath at higher lung volumes to produce the necessary after appropriate leak correction, showed a sensitivity and specificity in detecting EFL expiratory flow. To be effective, the PEEP level applied to the patient should be equal to PEEPi.

The continuous monitoring of EFL could be a useful tool to select the minimum PEEP level required to abolish it.

EFL can be detected using the forced oscillation technique (FOT) by an index which quantifies, for each breath, the within-breath variations of respiratory reactance (delta Xrs) at 5Hz.

ELIGIBILITY:
Inclusion Criteria

1. Age < 80 years
2. Moderate - Severe COPD diagnosed by spirometry (according to the GOLD criteria - Global Initiative for Chronic Obstructive Lung Disease criteria)
3. Free from any exacerbation in the 6 weeks preceding the study

Exclusion Criteria

1. Any co-existing cardio-pulmonary conditions which may result in a picture of ventilatory failure such as congestive cardiac failure, chest wall or neuromuscular disease, bronchopneumonia, pulmonary fibrosis, bronchiectasis, cystic fibrosis or obesity-hypoventilation syndrome
2. Clinically unstable; exacerbation within the preceding 6 weeks
3. The presence of pulmonary or extra-pulmonary neoplasia that is still active
4. The presence of a bleeding diathesis
5. Unstable coronary artery disease
6. Presence of tuberculosis, current infection or potentially infectious pathogen
7. Inability to provide informed consent to the study

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Calverley, Professor, Principal Investigator — Aintree University Hospital
Locations (1):
- University Hospital Aintree, Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and screened with spirometry and determination of expiratory flow limitation prior to being enrolled into the study.
Pre-assignment Details: 22 patient were recruited in June of 2010.
  * 13 patients studied
  * (7 didn't tolerate balloon; 2 had an exacerbation )
Groups:
- Therapy Arm: Non Invasive Ventilation using forced oscillation technique (FOT)
Period: Overall Study
Arm/Group | Therapy Arm
Started | 22
Completed | 13
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Therapy Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22

OUTCOME MEASURES:

1. Primary Outcome: Detection of Expiratory Flow Limitation
Description: Expiratory flow limitation (EFL) is an increase in transpulmonary pressure (cmH2O) with no change expiratory flow (lpm).
  Expiratory Flow Limitation or absence thereof will be detected by using a measurement of changes in reactance (DeltaXrs - cmH2O*s/L) it will be compared to the the Mead and Whittenberger technique (via esophageal balloon measuring transpulmonary pressures).
  Two measurements will be obtained, DeltaXrs and Transpulmonary pressure. Comparisons of these measurements will be made to determine if the participant exhibits EFL.
Time Frame: within 2 hours
Population: All participants that completed the protocol were analyzed.
Measure: Least Squares Mean (90% Confidence Interval); unit: cmH2O*s/L
Arm/Group | Therapy Arm
Number analyzed (Participants) | 13
cmH2O*s/L | 2.6 [2 to 3]
Statistical Analysis 1: Comparison: Therapy Arm; Test type: Other — Sensitivity and Specificity of values with respect to the Mead Whittenberger method were computed as follows (FL=flow limited and NFL = Non Flow limited): Sensitivity = (# of FL breaths detected by FOT / # of FL breaths detected by M&W) * 100 Specificity =(# of NFL breaths detected by FOT / # of NFL breaths detected by M&W) * 100; DeltaXrs (cmH2O*s/L) = 2.6, 90% CI 2-sided [0 to 100] — DeltaXrs equals average inspiratory reactance minus average expiratory reactance

2. Primary Outcome: Detection of Expiratory Flow Limitation by a Commercial Mechanical Ventilator
Description: Number of participants found to have expiratory flow limitation as determined by a commercial mechanical ventilator.
Time Frame: 2 hours
Population: All participants that completed the protocol were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy Arm
Number analyzed (Participants) | 13
Participants
  Flow limited | 8
  Not Flow Limited | 5

3. Primary Outcome: Detection of Expiratory Flow Limitation by Mead and Wittenberger (M-W) Technique
Description: Number of breaths are cumulative across all participants were found to be flow limited, not-flow limited or indeterminate as determined by the Mead and Wittenberger (M-W) technique of esophageal pressure. Each participant's individual breaths was imported into Matlab software program that displayed the flow vs transpleural pressure and breaths were individually analyzed according to the Mead Wittenberger technique.
Time Frame: 2 hours
Population: All participants that completed the protocol were analyzed.
Measure: Number; unit: breaths
Arm/Group | Therapy Arm
Number analyzed (Participants) | 13
breaths
  Flow limited | 534
  Not Flow Limited | 567
  Indeterminate | 1396

ADVERSE EVENTS:
Time Frame: Over course of the study which was 3 months in duration.
Arm/Group | Therapy Arm
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy Arm (N=22)
Chronic Obstructive Pulmonary Disease Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 2 participants had COPD exacerbations after consent but prior to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less